CLINICAL TRIAL: NCT05006651
Title: Video Laryngoscope vs. Video Stylet During General Anesthesia With Obesity Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB109-265-A
Record Dates: First submitted 2021-08-08; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Intubation; Difficult or Failed; Obesity
Keywords: obesity; Intubation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Laryngoscope (No Intervention): Intubation with traditional laryngoscope
- McGrath MAC (Active Comparator): Intubation with video laryngoscope
  Interventions: Device: McGrath MAC
- Trachway (Active Comparator): Intubation with video stylet
  Interventions: Device: Trachway

INTERVENTIONS:
Device: McGrath MAC — Intubaion with McGrath MAC
  Arms: McGrath MAC
Device: Trachway — Intubaion with Trachway
  Arms: Trachway

SUMMARY:
Obesity patients are more common in recent years. They have potential difficult airway. Two different video devices are popular used in Taiwan, video larygoscope and video stylet. We compared video larygoscope (McGrath MAC) and video stylet (Trachway) during elective surgery require tracheal intubation with obesity patients. The control group is traditional laryngoscope. 325 patients would be enrolled, above 100 patient each group.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery needs intubation
* ASA I to III
* BMI>30kg/m2

Exclusion Criteria:

* Head and neck cancer
* Skull, neck fracture
* Tracheal trauma
* NPO< 8hr
* Lung disease with hypoxemia
* Mental Disorders
* Patient wouldn't be extubated after operation immediately
* Contraindicated to muscle relaxant

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to Intubation | 10 minute
  Total intubation duration
Intubation difficulty | 10 minute
  Including Intubation difficulty scale, inubation attempt times, number of operator

SECONDARY OUTCOMES:
Any injury during intubation | 24 hours
  Including sore throat, hoarseness, trauma

CONTACTS AND LOCATIONS:
Overall Officials: Po-Kai Wang, Study Chair — Hualien Tzu Chi General Hospital
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Hualien, Taiwan

IPD SHARING:
Plan to Share IPD: No